CLINICAL TRIAL: NCT02977793
Title: Comparative Study of the TOMEY Specular Microscope EM-4000 and the Konan CellChek XL for the Measurements of Endothelial Cell Density, Coefficient of Variation of Endothelial Cell Area, % Hexagonality, Central Corneal Thickness
Brief Title: Comparative Study of the TOMEY Specular Microscope EM-4000 and the Konan CellChek XL
Status: Completed | Type: Observational
Sponsor: Tomey Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: TOMEY-EM4000-US-001
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Corneal and Endothelial Cell Measurements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Non-pathologic young adults: 18-28 years old
  Interventions: Device: Tomey EM-4000 Specular Microscope; Device: Konan CellChek XL Specular Microscope
- Non-pathologic adults: 29-80 years old
  Interventions: Device: Tomey EM-4000 Specular Microscope; Device: Konan CellChek XL Specular Microscope
- Pathologic adults: 29-80 years old
  Interventions: Device: Tomey EM-4000 Specular Microscope; Device: Konan CellChek XL Specular Microscope

INTERVENTIONS:
Device: Tomey EM-4000 Specular Microscope
Device: Konan CellChek XL Specular Microscope

SUMMARY:
The Tomey EM-4000 Specular Microscope is designed to observe and analyze corneal endothelium.

DETAILED DESCRIPTION:
The Tomey EM-4000 Specular Microscope is designed to observe and analyze corneal endothelium by capturing an image of corneal endothelium tissues. without making contact, analyzing the captured image, and calculating data such as cell density.

ELIGIBILITY:
Inclusion Criteria-Non-pathologic young adults (18-28 years old) and non-pathologic adults (29-80 years old)

1. Male or female subjects from 18 to 80 years old who have full legal capacity to volunteer on the date the informed consent is signed;
2. Subjects who can follow the instructions by the clinical staff at the clinical site, and can attend examinations on the scheduled examination date;
3. Subjects who agree to participate in the study.

Inclusion Criteria -Pathologic adults (29-80 years old):

1. Male and female subjects from 29 to 80 years old who have full legal capacity to volunteer on the date the informed consent is signed;
2. Subjects who can follow the instructions by the clinical staff at the clinical site, and can attend examinations on the scheduled examination date;
3. Subjects who agree to participate in the study;
4. At least one eye with any of the following conditions:

   1. History of post-op surgical trauma including pseudophakic or aphakic bullous keratopathy
   2. History of corneal transplant
   3. Physical injury or trauma to the cornea
   4. Fuch's dystrophy, Guttata or other corneal endothelial dystrophies
   5. Keratoconus
   6. Long-term polymethyl methacrylate (PMMA) contact lens use (greater than 3 years).

Exclusion Criteria - Non-pathologic young adults (18-28 years old) and non-pathologic adults (29-80 years old)

1. History of post-op surgical trauma including bullous keratopathy;
2. History of corneal transplant;
3. Evidence of physical injury or trauma to the cornea;
4. Fuch's dystrophy, Guttata or other corneal endothelial dystrophies;
5. Keratoconus;
6. Long-term PMMA contact lens use (greater than 3 years);
7. History of cataract, refractive or ocular surgical procedures that render the cornea opaque or otherwise impact its ability to be imaged using the investigational device;
8. Fixation problems which may prevent obtaining good Tomey EM-4000 and Konan CellChek XL images in either eye.

Exclusion Criteria - Pathologic adults (29-80 years old)

1. History of cataract, refractive or ocular surgical procedures that render the cornea opaque or otherwise impact its ability to be imaged using the investigational device;
2. Fixation problems which may prevent obtaining at least poor quality Tomey EM-4000 and Konan CellChek XL images in either eye.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects recruited can be male or female, of any race or ethnicity, ages 18-80 years of age at Visit 1. All subjects enrolled must meet all the inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Endothelial cell density measurements | 1 day
Coefficient of variation of endothelial cell area | 1 day
% Hexagonality | 1 day
Central Corneal Thickness | 1 day

SECONDARY OUTCOMES:
Adverse Events | 1 day

IPD SHARING:
Plan to Share IPD: No